CLINICAL TRIAL: NCT02268630
Title: Long Term Outcomes of Venous Thromboembolism -the LOVE Study-
Brief Title: Long Term Outcomes of Venous Thromboembolism
Acronym: LOVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LOVE1213
Record Dates: First submitted 2014-08-06; First posted 2014-10-20 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Post Thrombotic Syndrome; Chronic Thromboembolic Pulmonary Hypertension; Venous Thrombosis
Keywords: Post-thrombotic syndrome; Chronic thromboembolic pulmonary hypertension; Anticoagulation; Rivaroxaban
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: Patients treated with Warfarin for VTE
- Grup B: Patients treated with Rivaroxaban for VTE

SUMMARY:
This prospective observational follow-up study is designed to assess the long-term outcomes after Venous thromboembolism (VTE) and to assess the effect of the new oral anticoagulant (NOAC) rivaroxaban on the prevalence of post-thrombotic syndrome (PTS).

The study will not be testing any formal hypothesis.

DETAILED DESCRIPTION:
This prospective observational follow-up study is designed to assess the long-term outcomes after VTE and to assess the effect of NOAC (rivaroxaban) on the prevalence of PTS. All patients diagnosed and treated for VTE at SØF from 01.01.2011 will be invited to participate in this study. Newly diagnosed patients will be recruited and followed-up according to the study schedule which is based on state of the art international guidelines.

First follow-up will be performed at the end of treatment period, which is usually 3 or 6 months after an event of VTE, or at one year if patients will be put on permanent AC. Thereafter, patients will be followed-up annually for at least 5 years or up to the end of the study, i.e for 10 years.

The primary endpoints of the study are the development of PTS and CTEPH after VTE. There will be 3 visits: at 3 or 6 months depending on the duration of AC, at 2 and 5 years, in addition to a visit for TTE at 6 months. Remaining follow-ups will be performed by phone or by mail. All patients with PE will be examined by TTE 6 months after the diagnosis of PE. Those with signs of PAH will be referred for further work-up to establish the presence or absence of CTEPH at specialized centres. Patients with DVT will be evaluated for PTS at 2 and 5 years and for CTEPH if they develop dyspnoea. As for part b of the primary objective, the study will allow inclusion of patients with previous DVT diagnosed after 01.01.11.

ELIGIBILITY:
Inclusion Criteria:

* Patients with objectively verified first time DVT diagnosed after 01.01.11 for study A, OR objectively verified DVT and/or PE dignosed after 01.04.14 for study B.

  * 18 years of age
* Signed informed written consent

Exclusion Criteria:

* Patients who refuse to consent
* Patients who have been treated with other anticoagulants than thoose included in the study
* Patients who can not participate due to logistic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with VTE in Østfold who fulfil study criteria will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2014-01; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of post thrombotic syndrome and chronic thromboembolic pulmonary hypertension | 5 years
  Determine the prevalence of post thrombotic syndrome as defined by Villalta score at 2- and 5 years in an unselected population of venous thromboembolism patients.
  Prevalence of chronic thromboembolic pulmonary hypertension in at 2- and 5 years in an unselected population of pulmonary embolism patients.

SECONDARY OUTCOMES:
Bleeding | 9 years
  Rate of bleeding during treatment with anticoagulation
Recurrence rate | 9 years
  Recurrence rate during treatment and after discontinuation of anticoagulation.
Mortality rate | 9 years
  Mortality rate following deep vein thrombosis and /or pulmonary embolism.
Severity of pulmonary embolism | 9 years
  Severity of PE based on CT (Fredrikstad score) and troponin level.
Incidence of cancer | 9 years
  Incidence of cancer after diagnosis of venous tromboembolism in screened and unscreened patients
Compliance in the use of Elastic compression stockings | 9 years
  Compliance in the use of Elastic compression stockings
Risk factors | 9 years
  Risk factors for venous thromboembolism
Resource utilization | 9 years
  Resource utilization (number of contacts with health care providers, INR tests during anticoagulation)
Post thrombotic syndrome according to CEAP | 9 years
  PTS according to CEAP score

CONTACTS AND LOCATIONS:
Overall Officials: Kristin K Utne, MD, Principal Investigator — Ostfold Hospital Trust; Waleed Ghanima, PhD, Study Director — Ostfold Hospital Trust
Locations (3):
- Norway (3):
  - Akershus University Hospital, Lørenskog, Akershus
  - Ullevål University Hospital, Oslo, Oslo County
  - Ostfold Hospital Trust, Fredrikstad, Østfold fylke